CLINICAL TRIAL: NCT02064543
Title: Measurement of Gait Using the Opal APDM and an Instrumented Gait Mat in Persons With Parkinsonism
Brief Title: Measurement of Gait Using Opal APDM and Gait Mat in Parkinsonism
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 072012-090
Record Dates: First submitted 2014-01-22; First posted 2014-02-17 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Parkinsonism
Keywords: Parkinson's disease; gait
MeSH Terms: conditions — Parkinsonian Disorders; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ADPM and GAITRite: mobility assessments (ADPM, GAITRite) measuring gait parameters
  Interventions: Other: GAITRite; Other: ADPM

INTERVENTIONS:
Other: GAITRite — mobility test assessing gait parameters
Other: ADPM — mobility test assessing gait parameters

SUMMARY:
The project is a prospective trial comparing Zeno/GAITRite and APDM® in a cohort of persons living with parkinsonian disorders. Ambulatory patients with a parkinsonian syndrome and who are able to provide informed consent will participate in the assessments.

Outcome variables include selected gait and balance parameters such as cadence, gait-cycle, stride-length, stride-velocity, turning duration, turning steps, postural sway and anticipatory postural control. These parameters will be measured by the portable inertial sensors developed by APDM® and the Zeno/GaitRite.

DETAILED DESCRIPTION:
Testing

Participants after screening and consenting will:

1. Have their height measured and fit with the APDM Opals (each device is a two inch square attached by velcro), one device is attached to each leg, each arm, and the trunk and chest and receive an introduction to walking on the gait mat.
2. Participants are then asked to walk at a self selected walking speed down the gait mat. The participants will complete multiple passes (8-10 passes, total 75-100 feet) across the gait mat while wearing the APDM units to concurrently collect all temporal and spatial data needed to answer the research question. The Zeno mat is the intended primary gait mat for this study. The GaitRite will only be utilized in the case of a technical issue with the Zeno in order to insure completion of the data collection.

ELIGIBILITY:
Inclusion Criteria

1. Adults between the ages of 18 and 80 years of age with a primary diagnosis of PD and similar parkinsonian syndromes
2. Individuals able to walk 100 feet independently, with or without the use of an assistive device (walker, cane) and follow simple instructions.
3. Individuals with sufficient physiological systemic support to participate in the study protocol

Exclusion Criteria

1. Inability to speak English secondary to the need to understand and follow multistep directions
2. A secondary diagnosis (musculoskeletal, cardiopulmonary, neurological) that excludes participation in the study
3. Inability to ambulate 100 feet independently with or without an assistive device.
4. Inability to follow simple instructions necessary for completion of the testing tasks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between the ages of 18 and 80 years of age with a primary diagnosis of PD and similar parkinsonian syndromes and clinical signs of FoG
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
gait parameters | one year
  Outcome variables include selected gait and balance such as cadence
gait parameters | one year
  Outcome variables include selected gait and balance such as stride-length
gait parameters | one year
  Outcome variables include selected gait and balance such as stride-velocity
gait parameters | one year
  Outcome variables include selected gait and balance such as turning duration
gait parameters | one year
  Outcome variables include selected gait and balance such as turning steps
gait parameters | one year
  Outcome variables include selected gait and balance such as postural sway
gait parameters | one year
  Outcome variables include selected gait and balance such as anticipatory postural control

CONTACTS AND LOCATIONS:
Overall Officials: Pravin Khemani, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No